CLINICAL TRIAL: NCT00153426
Title: West Virginia WISEWOMAN Project
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: West Virginia University (Other)
Responsible Party: Principal Investigator, Robin Seabury, Associate Director, West Virginia University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: CDC-NCCDPHP-4234; U58/CCU322798-01
Record Dates: First submitted 2005-09-08; First posted 2005-09-12 (Estimated); Last update posted 2012-06-28 (Estimated); Status verified 2012-06

CONDITIONS: Risk Reduction Behavior
MeSH Terms: conditions — Risk Reduction Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- lifestyle counseling (Experimental): Women assigned to lifestyle change intervention arm for nutrition and physical activity with print-based tailored health communications and a computer-based interactive nutrition program targeting health behaviors of diet and physical activity. Women in a control group did not receive the intervention.
  Interventions: Behavioral: West Virginia WISEWOMAN

INTERVENTIONS:
Behavioral: West Virginia WISEWOMAN — Print-based tailored health communications and computer-based interactive nutrition program

SUMMARY:
To provide low-income, under- or uninsured 40- to 64-year-old women with the knowledge, skills, and opportunities to improve diet, physical activity, and other lifestyle behaviors to prevent, delay and control cardiovascular and other chronic diseases.

ELIGIBILITY:
Inclusion Criteria:

* NBCCEDP

Exclusion Criteria:

-

Ages: 40 Years to 64 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 733 (Actual)
Dates: Start 2003-07; Primary Completion 2008-03 (Actual); Study Completion 2008-03 (Actual)

PRIMARY OUTCOMES:
change in physical activity and nutrition lifestyle behaviors | baseline and one year

CONTACTS AND LOCATIONS:
Overall Officials: Julie Will, Study Chair — Centers for Disease Control and Prevention